CLINICAL TRIAL: NCT07113535
Title: RAM Cannula Versus Short Binasal Prong Interfaces of Non- Invasive Ventilation for Prevention of Extubating Failure in Preterm Infants: A Randomized Controlled Trial
Brief Title: Post-extubation Use RAM Cannula Versus Short Binasal Prong Interfaces in Preterm Infants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, hussam murayh mohammed ali, Fellow of Neonatal- perinatal medicine, NICU, Ministry of Health, Saudi Arabia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-03-M-11
Record Dates: First submitted 2025-07-28; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Premature; Respiratory Distress Syndrome; Extubation
Keywords: nasal interface; noninvasive respiratory support; premature; RAM cannula; Chest ultrasound; Diaphragm
MeSH Terms: conditions — Premature Birth; Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RAM cannula group (Active Comparator): Preterm infants will receive non-invasive ventilation by RAM cannula
  Interventions: Other: RAM cannula
- Short binasal prong group (Active Comparator): Preterm infants will receive non-invasive ventilation by short binasal prongs
  Interventions: Other: Short binasal prong

INTERVENTIONS:
Other: RAM cannula — RAM cannula as an interface for non invasive ventilation in preterm newborns
  Arms: RAM cannula group
Other: Short binasal prong — Short binasal prong as an interface for non invasive ventilation in preterm newborns
  Arms: Short binasal prong group

SUMMARY:
Nowadays, the use of non-invasive ventilation for preterm infants in the NICU has increased to avoid complications associated with prolonged endotracheal intubation. Adequate pressure delivery through non-invasive ventilation is essential, as it enhances the growth and development of premature lungs. Various interfaces have been used to ensure proper sealing. The RAM cannula, used as an interface for non-invasive respiratory support in preterm neonates, is associated with reduced nasal trauma compared to short binasal prongs (SBPs), due to its softer material, making it a safer option. However, the RAM cannula has been shown to deliver lower pharyngeal pressure and, therefore, may not maintain airway pressure as consistently as nasal prongs. Currently, limited data is available regarding the efficacy of nasal prongs compared to the RAM cannula as a post-extubation interface for non-invasive ventilation support in preterm infants. Additionally, we have observed that the use of the RAM cannula for non-invasive ventilation in preterm infants is associated with a longer duration of oxygen therapy compared to SBPs.

The investigators hypothesize that the RAM cannula provides a lower level of positive end-expiratory pressure compared to SBPs during non-invasive ventilation.

The investigators aim to assess the efficacy and safety of the RAM cannula versus SBPs as nasal interfaces for post-extubation non-invasive respiratory support in preterm infants.

DETAILED DESCRIPTION:
Preterm infants will be randomized to receive post-extubation non invasive respiratory support either through RAM cannula or SBPs. Neonates in both groups will be uniformly managed as per unit protocol as following:

Extubation criteria :

* Birth weight < 1000 gram :MAP <7 cmH2O and FIO2 <0.30
* Birth weight>1000 gram :MAP >8 cmH2O and FIO2 <0.30

Re intubation criteria :

* FIO2>0.60 to maintain SaO2 >88% OR PaO2 > 45 mmHg
* PaCO2 {arterial} > 55-60 with PH < 7.25
* Apnea and requiring bag and mask ventilation
* Evidence of increased work of breathing {retractions -grunting -chest wall distortion } plus abnormal chest x ray

ELIGIBILITY:
Inclusion Criteria:

* Inborn preterm neonates ≤ 32 weeks of gestational and/or birth weight ≤1500 g with respiratory distress syndrome requiring initial invasive ventilation support for at least 24 hours.

Exclusion Criteria:

* Outborn preterm neonates
* Major congenital malformations.

Ages: 24 Hours to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Failure of extubation incidence rate | 28 days of an infant's life
  Need for reintubation within 72 hours post-extubation trial

SECONDARY OUTCOMES:
Duration of non-invasive ventilation | 120 days
  Days on non-invasive ventilation
whole duration of oxygen therapy | 120 days
  Days on oxygen therapy during NICU admission
Diaphragmatic indices and lung ultrasound scores post-extubation (pre & post extubation then weekly) | 120 days
  Diaphragmatic indices (diaphragmatic thickness &excursion) and lung ultrasound scores post-extubation
Need for reintubation within 7 days | 28 days of an infant's life
  Need for reintubation within 72 hours post-extubation trial
Bronchopulmonary dysplasia | 120 days
Mortality | 120 days
  Pre-discharge mortality

CONTACTS AND LOCATIONS:
Overall Officials: Nehad Nasef, Dr, Principal Investigator — King Salman Bin Abdulaziz Medical City
Locations (1):
- King Salman Bin Abdulaziz Medical City, Madinah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers for research and scientific purposes (i.e conduction of meta-analysis or systematic review). Data or samples shared will be coded, with no protected health information included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol
Time Frame: Data requests can be submitted starting 3 months after article publication and the data will be made accessible for up to 12 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to raw data (no protected health information) can be requested by qualified researchers for scientific purposes, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA)

REFERENCES:
- [Background] Gokce IK, Kaya H, Ozdemir R. A randomized trial comparing the short binasal prong to the RAM cannula for noninvasive ventilation support of preterm infants with respiratory distress syndrome. J Matern Fetal Neonatal Med. 2021 Jun;34(12):1868-1874. doi: 10.1080/14767058.2019.1651268. Epub 2019 Aug 8. PMID 31394948